CLINICAL TRIAL: NCT01670292
Title: Patient Response to Spinal Manipulation
Acronym: PRiSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: University of Iowa (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRiSM Study; U19AT004663 (NIH)
Record Dates: First submitted 2012-08-02; First posted 2012-08-22 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: HVLA-SM (Other): Experimental High Velocity Low Amplitude Spinal Manipulation
  Interventions: Other: HVLA-SM

INTERVENTIONS:
Other: HVLA-SM — High Velocity Low Amplitude Spinal Manipulation

SUMMARY:
This is a biomechanical study which is Project 1 in the Developmental Center for Clinical and Translational Research in Chiropractic (DCRC I) (NIH/NCCAM grant 1 U19 AT004663-01; principal investigator Christine Goertz, DC, PhD). This study is designed to monitor both physiological and patient self-report outcome variables. In addition, as there is little quantitative information on Spinal Manipulation Technique procedures reported in clinical trials, the study is designed to collect preliminary kinetic measures of the spinal manipulation technique delivery (i.e. force-time profiles).

DETAILED DESCRIPTION:
Participants with narrowly defined chronic low back pain will be included in this study. Each participant will be treated 12 times over the course of 6 weeks. The following data will be collected: participant characteristics that may predict outcome or be modifiers of force used by provider (gender, age, height, weight, and Body Mass Index); spinal segment load during the pre-load and thrusting phases (force and moment in the pre-load phase, peak load, and loading rate); physiological measures (posterior-anterior global stiffness and flexion-relaxation); patient-centered outcomes of back pain and function; and adverse events.

Study participants (n= 80) will be recruited from the Quad Cities metro area. A team of experienced chiropractic clinicians working at the Palmer Center for Chiropractic Research will treat study participants. Each of the study participants will receive 2 High Velocity Low Amplitude Spinal Manipulation treatment visits per week over a 6 week period. The physiological assessments will be performed immediately before and after Spinal Manipulation delivery during treatment visits 1, 5 & 12 (6 sets of assessments in total). During these same treatment visits, we will also capture the kinetic measures during Spinal Manipulation delivery for spinal segment load analysis. Participant patient-centered outcomes will be measured at baseline 1, and treatment visits 6 and 13. For simplicity, data collection time points will be named as baseline, after 2 weeks, and after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* NRS score, AVERAGE within the past 24 hours
* Must be ≥4 at the phone screen or baseline 1 visit
* Must be ≥2 at phone screen, baseline 1 and baseline 2 visits
* Roland Morris Disability ≥6
* Age 21-65
* Signed informed consent document
* Chronic (12+ weeks) low back pain

Exclusion Criteria:

* Compliance concerns
* No manipulable lesion in L1-L5 or SI joints
* The absence of typical palpatory characteristics as well as the absence of a global assessment that would indicate that spinal manipulation is likely to generate a positive therapeutic effect, even without the presence of standard palpatory findings
* Ongoing treatment for low back pain by outside provider
* Comorbid conditions
* Serious concomitant illness
* Inflammatory or destructive spinal tissue change
* Ankylosing Spondylytis
* Fibromyalgia
* Rheumatoid Arthritis
* Confirmed or suspected disc herniation with neurological signs
* Neuromuscular disease (e.g. Parkinson's, Muscular Dystrophy, Cerebral Palsy, or Myasthenia gravis
* Spinal surgery <6 months
* Suspicion of drug or alcohol dependence or abuse
* Uncontrolled hypertension
* Lower extremity peripheral arterial disease
* Undetermined, infections or visceral source of low back pain
* Other comorbid conditions prohibiting treatment and/or testing
* Safety concerns
* Bleeding disorders
* Contraindications to High Velocity Low Amplitude Spinal Manipulation
* Inability to tolerate or obtain positon for flexion-relaxation test without condition aggravation
* Inability to tolerate or perform/receive any study procedure without condition aggravation
* Quebec Task Force (QTF) criterion 4-11:
* QTF 4: Pain + radiation to upper/lower limb with neurologic signs
* QTF 5: Presumptive compression of a spinal nerve root on a simple roentgenogram
* QTF 6: Compression of a spinal nerve root confirmed by specific imaging techniques
* QTF 7: Spinal Stenosis
* QTF 8: Postsurgical status, 1-6 months after intervention
* QTF 9: Postsurgical status, >6 months after intervention
* QTF 10: Chronic pain syndrome
* QTF 11: Other diagnoses
* Pregnancy
* Pacemaker or defibrillator
* Inability to read or verbally comprehend English
* Joint replacement
* Use of spinal manipulation within past 4 weeks
* Sensitivity to adhesive
* Diagnostic procedures other than x-ray/UA necessary
* BDI-II ≥29
* Retention of legal advice and open or pending case related to low back pain
* BMI ≥40
* Unwilling to have low back and wrist shaved
* Moving from Quad Cities area within next 8 weeks
* Unwilling to postpone treatments for low back pain from another provider
* Seeking or receiving compensation for any disability

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Xia, PhD, Principal Investigator — Palmer College of Chiropractic
Locations (1):
- Palmer College of Chiropractic, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the resulting manuscripts have been published, data sets will be provided for public access. Potential investigators can contact one of the Co-PIs to present their hypothesis, study design, instruments and/or data on which to focus, and resources required. Depending upon the needs and desires of the requesting party, the data that are shared may include analytic tables or de-identified or limited data sets that are transmitted to the requesting parties for additional analyses.

REFERENCES:
- [Background] Xia T, Wilder DG, Gudavalli MR, DeVocht JW, Vining RD, Pohlman KA, Kawchuk GN, Long CR, Goertz CM. Study protocol for patient response to spinal manipulation - a prospective observational clinical trial on physiological and patient-centered outcomes in patients with chronic low back pain. BMC Complement Altern Med. 2014 Aug 8;14:292. doi: 10.1186/1472-6882-14-292. PMID 25106673
- [Background] Minkalis AL, Vining RD. What is the pain source? A case report of a patient with low back pain and bilateral hip osteonecrosis. J Can Chiropr Assoc. 2015 Sep;59(3):300-10. PMID 26500365
- [Derived] Xia T, Long CR, Vining RD, Gudavalli MR, DeVocht JW, Kawchuk GN, Wilder DG, Goertz CM. Association of lumbar spine stiffness and flexion-relaxation phenomenon with patient-reported outcomes in adults with chronic low back pain - a single-arm clinical trial investigating the effects of thrust spinal manipulation. BMC Complement Altern Med. 2017 Jun 9;17(1):303. doi: 10.1186/s12906-017-1821-1. PMID 28599647
- See also: Study protocol for patient response to spinal manipulation - a prospective observational clinical trial on physiological and patient-centered outcomes in patients with chronic low back pain — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4139615/
- See also: What is the pain source? A case report of a patient with low back pain and bilateral hip osteonecrosis. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4593036/

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: HVLA-SM: Experimental High Velocity Low Amplitude Spinal Manipulation
  HVLA-SM: High Velocity Low Amplitude Spinal Manipulation
  Participants receive treatments of HVLA-SM to the lumbar spine in the side-lying position. Treatment frequency is twice per week for 6 weeks.
Period: Overall Study
Arm/Group | Experimental: HVLA-SM
Started | 82
Completed | 68
Not Completed | 14
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: HVLA-SM
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 43
Baseline Patient-Centered Outcome Measures [Mean (Standard Deviation); unit: units on a scale] — VAS - Visual Analog Scale: The VAS is a single-item, unidimensional measure for pain. Score interpretations for the VAS include the following cut points: no pain (0 to 4 mm), mild pain (5 to 44 mm), moderate pain (45 to 74 mm), and severe pain (75 to 100 mm).
  RMDQ - Roland Morris disability questionnaire: The RMDQ consists of 24 questions related to disability, with each question worth one point. Scores can range from 0 (no disability) to 24 (severe disability).
  units on a scale
    VAS | 46.1 (18.1)
    RMDQ | 9.5 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Patient-Centered Outcome Measurement Mean Change After 6 Weeks (VAS, RMDQ)
Description: VAS - Visual Analog Scale - Scale: 0-100 mm (anchors: 0 mm = No Pain, 100 mm = Worst Imaginable Pain). VAS Interpretation: A higher score indicates greater pain intensity. In this study, improvement of 30% from the baseline value was considered clinically significant.
  RMDQ - Roland Morris disability questionnaire - Scale: 0 (no disability) to 24 (maximum disability). RMDQ Interpretation: Greater levels of disability are reflected by higher scores. In this study, improvement of 30% from the baseline value was considered clinically significant.
Time Frame: Baseline to 6 weeks
Population: 82 and 68 participants completed at baseline and after 6 weeks, respectively. Data from all participants (n=82) were used in statistical analysis. The reported data represents the mean change from baseline to week 6.
Measure: Mean (95% Confidence Interval); unit: units on a scale (see description above)
Arm/Group | Experimental: HVLA-SM
Number analyzed (Participants) | 82
units on a scale (see description above)
  Mean Reduction in VAS score (mm) | 20.1 [14.1 to 26.1]
  Mean Reduction in RMDQ score | 4.8 [3.7 to 5.8]

2. Primary Outcome: Lumbar-spine Stiffness (LSS)
Description: LSS* contains 5 variables: global stiffness (GS, unit: Newton/mm) at L3 from 1) hand palpation 2) a hand-held device & 3) an automated indenter device; global stiffness variation (GSV, unit: Newton/mm) between GS from L1 to L5 from 4) hand palpation & 5) a hand-held device.
  *LSS Interpretation: The values of the outcome depend on testing procedure, instruction to participants, and equipment. Currently there is no consensus regarding what value is high than normal, normal, lower than normal.
Time Frame: Baseline, 2 weeks, 6 weeks
Population: 82, 71 and 68 participants completed at baseline, after 2 weeks and after 6 weeks, respectively. The number of observations at each of the 3 time points for individual measures is equal to or lower than these numbers due to missing data.
Measure: Mean (Standard Deviation); unit: N/mm
Groups:
- HVLA-SM at Baseline: Results at Baseline
  Experimental High Velocity Low Amplitude Spinal Manipulation
  HVLA-SM: High Velocity Low Amplitude Spinal Manipulation
- HVLA-SM After 2 Weeks: There is only one group/arm, this is the data for the same group of participants after two weeks.
- HVLA-SM After 6 Weeks: There is only one group/arm, this is the data for the same group of participants after six weeks.
Arm/Group | HVLA-SM at Baseline | HVLA-SM After 2 Weeks | HVLA-SM After 6 Weeks
Number analyzed (Participants) | 82 | 71 | 68
N/mm
  LSS - Palpatory - GS (N/mm) at L3 | 4.8 (1.8) | 4.3 (1.8) | 4.2 (1.3)
  LSS - Hand-held - GS (N/mm) at L3 | 7.7 (2.1) | 7.5 (1.8) | 7.6 (2.2)
  LSS - Automated - GS (N/mm) at Ant | 5.2 (1.5) | 5.3 (1.4) | 5.3 (1.5)
  LSS - Palpatory - GSV (N/mm) | 2.3 (1.5) | 2.0 (1.1) | 1.9 (1.1)
  LSS - Hand-held - GSV (N/mm) | 2.3 (1.3) | 2.1 (1.1) | 2.1 (1.3)

3. Primary Outcome: Lumbar-spine Stiffness (LSS) - Normalized Global Stiffness Variation
Description: LSS contains 2 variables: Palpatory and Handheld device - normalized global stiffness variation (nGSV, unitless).
  LSS Interpretation: The values of the outcome depend on testing procedure, instruction to participants, and equipment. Currently there is no consensus regarding what value is higher than normal, normal, lower than normal.
Time Frame: Baseline, 2 weeks, 6 weeks
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | HVLA-SM at Baseline | HVLA-SM After 2 Weeks | HVLA-SM After 6 Weeks
Number analyzed (Participants) | 82 | 71 | 68
unitless
  LSS - Palpatory - nGSV | 0.5 (0.2) | 0.5 (0.2) | 0.5 (0.2)
  LSS - Hand-held - nGSV | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.1)

4. Primary Outcome: Flexion-Relaxation Ratio (FRR)
Description: FRR contains 4 variables, which are the average right and left back muscle FRR obtained using 1) maximum EMG during flexion, and 2) maximum EMG during extension to normalize EMG during full flexion; and asymmetry between the right and left back muscle FRRs using 3) maximum EMG during flexion, and 4) maximum EMG during extension to normalize EMG during full flexion
  FRR Interpretation: The values of the outcome depend on testing procedure, instruction to participants, and equipment. Currently there is no consensus regarding what value is high than normal, normal, lower than normal.
Time Frame: Baseline, 2 weeks, 6 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HVLA-SM at Baseline | HVLA-SM After 2 Weeks | HVLA-SM After 6 Weeks
Number analyzed (Participants) | 82 | 71 | 68
ratio
  Flexion FRR | 4.7 (3.7) | 5.8 (5.4) | 5.5 (5.6)
  Extension FRR | 9.2 (9.5) | 10.4 (11.6) | 9.4 (10.5)
  Asymmetry in flexion FRR | 1.5 (0.5) | 1.4 (0.5) | 1.4 (0.4)
  Asymmetry in extension FRR | 1.4 (0.7) | 1.4 (0.4) | 1.4 (0.5)

5. Secondary Outcome: Kinetic Measure - Spinal Segment Load (SSL) Force
Description: SSL* contains variables: maximum amplitude (Newton) during preload and peak thrust force in anterior-posterior (X), side-to-side (Y), head-to-toe direction (Z) and combined force (C).
  *Interpretation: the purpose of the outcomes is to quantify force-time profile of SM. The values of the outcome depend on the doctor who delivers SM, location and direction of SM, participant body position, and equipment. Currently there is no consensus regarding what value is higher than normal, normal, or lower than normal.
  Sign convention: because patient position would affect the sign of some measurements, the right side up position was used as the reference position (i.e., the affected measurements assessed in the left side up position had their sign inverted) in order to calculate mean and SD. The value reported is the change from baseline to week 6.
Time Frame: 6 weeks
Population: Note: 82, 71 and 68 participants completed at baseline, after 2 weeks and after 6 weeks, respectively, and a total of 593 SM was delivered during visits 1, 5, and 12. The number of observations for individual measures is lower than the total number of analyzable SM (n=575) due to missing data in corresponding components.
Measure: Mean (Standard Deviation); unit: Newton (N)
Units Other Than Participants: Spinal Manipulations
Groups:
- Anterior-Posterior (X): All participants are in this group, this simply defines the mean force/moment in the X direction.
- Side-to-Side (Y): All participants are in this group, this simply defines the mean force/moment in the Y direction.
- Head-to-Toe (Z): All participants are in this group, this simply defines the mean force/moment in the Z direction.
- Combined: All participants are in this group, this simply defines the mean Combined force/moment (C).
Arm/Group | Anterior-Posterior (X) | Side-to-Side (Y) | Head-to-Toe (Z) | Combined
Number analyzed (Participants) | 68 | 68 | 68 | 68
Number analyzed (Spinal Manipulations) | 575 | 575 | 575 | 575
Newton (N)
  Preload force (N) | -56.5 (87.2) | -67.0 (55.0) | -117.2 (59.4) | 170.3 (64.9)
  Peak thrust force (N) | -128.3 (163.4) | -172.3 (141.9) | -276.4 (137.1) | 385.1 (169.5)

6. Secondary Outcome: Kinetic Measure - Spinal Segment Load (SSL) Moment
Description: SSL* contains variables: maximum amplitude (Newton*Meter for moment) during preload and peak thrust force in anterior-posterior (X), side-to-side (Y), head-to-toe direction (Z) and combined force (C).
  *Interpretation: the purpose of the outcomes is to quantify force-time profile of SM. The values of the outcome depend on the doctor who delivers SM, location and direction of SM, participant body position, and equipment. Currently there is no consensus regarding what value is higher than normal, normal, or lower than normal.
  Sign convention: because patient position would affect the sign of some measurements, the right side up position was used as the reference position (i.e., the affected measurements assessed in the left side up position had their sign inverted) in order to calculate mean and SD. The value reported is the change from baseline to week 6.
Time Frame: 6 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Newton*Meter
Units Other Than Participants: Spinal Manipulations
Arm/Group | Anterior-Posterior (X) | Side-to-Side (Y) | Head-to-Toe (Z) | Combined
Number analyzed (Participants) | 68 | 68 | 68 | 68
Number analyzed (Spinal Manipulations) | 575 | 575 | 575 | 575
Newton*Meter
  Preload moment (N*M) | 19.8 (23.4) | -1.0 (19.4) | -45.4 (29.4) | 58.5 (27.8)
  Peak thrust moment (N*M) | 31.0 (46.0) | -3.4 (39.9) | -76.0 (42.2) | 99.5 (41.9)

7. Secondary Outcome: Kinetic Measure - Spinal Segment Load (SSL) Rate of Loading for Force
Description: SSL* contains variables: rate of loading for force in anterior-posterior (X), side-to-side (Y), head-to-toe direction (Z) and combined force (C).
  *Interpretation: the purpose of the outcomes is to quantify force-time profile of SM. The values of the outcome depend on the doctor who delivers SM, location and direction of SM, participant body position, and equipment. Currently there is no consensus regarding what value is higher than normal, normal, or lower than normal.
  Sign convention: because patient position would affect the sign of some measurements, the right side up position was used as the reference position (i.e., the affected measurements assessed in the left side up position had their sign inverted) in order to calculate mean and SD. The value reported is the change from baseline to week 6.
Time Frame: 6 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Newton/second
Units Other Than Participants: Spinal Manipulations
Arm/Group | Anterior-Posterior (X) | Side-to-Side (Y) | Head-to-Toe (Z) | Combined
Number analyzed (Participants) | 68 | 68 | 68 | 68
Number analyzed (Spinal Manipulations) | 575 | 575 | 575 | 575
Newton/second | -599.2 (897.1) | -598.1 (668.8) | -1145.2 (713.6) | 1537.5 (955.4)

8. Secondary Outcome: Kinetic Measure - Spinal Segment Load (SSL) Rate of Loading for Moment
Description: SSL* contains variables: rate of loading for moment in anterior-posterior (X), side-to-side (Y), head-to-toe direction (Z) and combined force (C).
  *Interpretation: the purpose of the outcomes is to quantify force-time profile of SM. The values of the outcome depend on the doctor who delivers SM, location and direction of SM, participant body position, and equipment. Currently there is no consensus regarding what value is higher than normal, normal, or lower than normal.
  Sign convention: because patient position would affect the sign of some measurements, the right side up position was used as the reference position (i.e., the affected measurements assessed in the left side up position had their sign inverted) in order to calculate mean and SD. The value reported is the change from baseline to week 6.
Time Frame: 6 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Newton*Meters/second
Units Other Than Participants: Spinal Manipulations
Arm/Group | Anterior-Posterior (X) | Side-to-Side (Y) | Head-to-Toe (Z) | Combined
Number analyzed (Participants) | 68 | 68 | 68 | 68
Number analyzed (Spinal Manipulations) | 575 | 575 | 575 | 575
Newton*Meters/second | 51.3 (201.8) | -40.4 (183.7) | -210.2 (159.0) | 275.2 (194.9)

9. Secondary Outcome: PROMIS-29 - Patient Reported Outcomes Measurement Information Scale-29: General Health Status Scale
Description: 1) The questionnaire contains 7 PROMIS-29 specific items: Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction with Participation in Social Role (anchors: 1= 'Not at all', 5= 'Very much', higher score is worse).
  Each PROMIS-29 specific item is reported in raw score (4-20) and scored in T-score (T), which rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10 for a population.
  On the T-score metric & interpretation:
  * A score of 40 is one SD lower than the mean of the reference population.
  * A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
Time Frame: Baseline, 2 weeks, 6 weeks
Population: Note: 82, 71 and 68 participants completed at baseline, after 2 weeks and after 6 weeks, respectively. Number of observations made at the three time points were 82, 70, and 68, respectively.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- HVLA-SM at Baseline: Result at baseline. Experimental High Velocity Low Amplitude Spinal Manipulation
  HVLA-SM: High Velocity Low Amplitude Spinal Manipulation
Arm/Group | HVLA-SM at Baseline | HVLA-SM After 2 Weeks | HVLA-SM After 6 Weeks
Number analyzed (Participants) | 82 | 70 | 68
T-score
  P29 - Anxiety | 49.18 (8.87) | 47.93 (7.87) | 46.58 (7.78)
  P29 - Depression | 47.02 (7.78) | 45.97 (7.07) | 44.38 (6.06)
  P29 - Fatigue | 53.72 (8.19) | 51.93 (7.84) | 50.09 (7.87)
  P-29 - Pain Interference | 60.26 (5.70) | 57.78 (6.37) | 55.12 (7.52)
  P29 - Physical Function | 33.31 (3.93) | 32.29 (3.84) | 30.07 (3.97)
  P29- Sleep Disturbance | 52.23 (3.13) | 51.11 (3.23) | 51.79 (3.10)
  P29 - Satisfaction w/ Participation in Social Role | 45.45 (6.84) | 46.51 (6.75) | 49.75 (7.71)

10. Secondary Outcome: PROMIS-29 - Patient Reported Outcomes Measurement Information Scale-29: Global Item, Pain NRS
Description: 1) The PROMIS questionnaire contains 1 PROMIS global item: Pain NRS, Scale: 0-10 (anchors: 0 = No Pain, 10 = Worst Imaginable Pain, higher score is worse). The PROMIS global item is not scored but reported in raw score.
Time Frame: Baseline, 2 weeks, 6 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HVLA-SM at Baseline | HVLA-SM After 2 Weeks | HVLA-SM After 6 Weeks
Number analyzed (Participants) | 82 | 70 | 68
units on a scale | 5.57 (1.63) | 4.46 (1.95) | 3.59 (2.18)

11. Secondary Outcome: Bothersomeness
Description: Question asked of participants: "During the past week, how bothersome have each of the following symptoms been?" The bothersomeness questionnaire contains two items: a) low back pain & b) leg pain (sciatica).
  Scale: 0-10 (anchors: 0 = Not at all bothersome, 10 = Extremely bothersome)
Time Frame: Baseline, 2 weeks, 6 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HVLA-SM at Baseline | HVLA-SM After 2 Weeks | HVLA-SM After 6 Weeks
Number analyzed (Participants) | 82 | 70 | 68
units on a scale
  Low Back Pain | 6.18 (1.93) | 4.80 (2.14) | 3.63 (2.30)
  Leg Pain (Sciatica) | 3.29 (3.18) | 2.61 (2.91) | 1.94 (2.68)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Any untoward medical occurrence that may present itself during the conduct of the study which may or may not have a causal relationship with the study procedures.
  *The total number of AEs may exceed the total # of people affected because some people experienced multiple AEs.
Groups:
- Experimental: HVLA-SM*: Experimental High Velocity Low Amplitude Spinal Manipulation
  HVLA-SM: High Velocity Low Amplitude Spinal Manipulation
Arm/Group | Experimental: HVLA-SM*
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 74/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: HVLA-SM* (N=82)
Neck pain/stiffness (Musculoskeletal and connective tissue disorders) | 2
Low back pain/stiffness (Musculoskeletal and connective tissue disorders) | 29
Neck and back pain/stiffness (Musculoskeletal and connective tissue disorders) | 2
Headache and neck/back pain (Musculoskeletal and connective tissue disorders) | 2
Back pain and extremity pain/stiffness (Musculoskeletal and connective tissue disorders) | 20
Thoracic and low back pain/stiffness (Musculoskeletal and connective tissue disorders) | 5
Neck, back and extremity pain/stiffness (Musculoskeletal and connective tissue disorders) | 4
Back and extremity pain/stiffness (Musculoskeletal and connective tissue disorders) | 2
Neck and extremity pain/stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain/stiffness in the extremities (Musculoskeletal and connective tissue disorders) | 1
Lower/extremity pain/stiffness (Musculoskeletal and connective tissue disorders) | 2
Neck and back pain and extremity pain and headache (Musculoskeletal and connective tissue disorders) | 1
Back pain/stiffness and numbness/tingling (Musculoskeletal and connective tissue disorders) | 1
Back pain and extremity pain and numbness/tingling (Musculoskeletal and connective tissue disorders) | 1
Upper respiratory infection (General disorders) | 5
Sinus congestion/upper respiratory symptoms/allergy (General disorders) | 5
Insect bite (General disorders) | 1
Hypertension (General disorders) | 1
Gastrointestinal symptoms (General disorders) | 1
Hemorrhoids (General disorders) | 1
Nausea and tooth/facial pain and sinus congestion (General disorders) | 1
Nausea and back pain/stiffness (General disorders) | 1
Dental caries (General disorders) | 1
Asthma and lower respiratory infection (General disorders) | 1
Upper respiratory infection and allergy (General disorders) | 1
Hemorrhoids and nasal congestion (General disorders) | 1
Laceration (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes